CLINICAL TRIAL: NCT01758484
Title: FEASIBILITY OF IMPLEMENTING PRE-TRANSPLANT EVALUATION BY THE SUPPORTIVE CARE TEAM FOR PATIENTS UNDERGOING HEMATOPOIETIC CELL TRANSPLANTATION FOR HEMATOLOGICAL MALIGNANCIES
Brief Title: Supportive Care for Patients With Hematological Malignancies Undergoing Hematopoietic Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2659.00; NCI-2012-03009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Hematopoietic/Lymphoid Cancer
Keywords: Hematopoietic cell transplantation; Supportive/palliative care
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (palliative care support) (Experimental): Patients undergo palliative care support before transplantation and at least once monthly while they remain at the transplant center.
  Interventions: Other: palliative care; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: palliative care — Undergo supportive care intervention
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies supportive care for patients with hematological malignancies undergoing hematopoietic cell transplant. Supportive care may improve quality of life in this patient population.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Pilot a supportive care intervention that begins prior to transplantation and continues through the acute peritransplant period.

II. Determine the proportion of patients who enroll and the level of comfort / distress of hematopoietic cell transplant (HCT) patients who meet with the supportive care team.

III. Pilot data collection mechanisms and cost retrieval in preparation for a randomized clinical trial.

OUTLINE:

Patients undergo supportive care consultation before transplantation and at least once monthly while they remain at the transplant center.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* English as primary language
* Planned autologous or allogeneic hematopoietic cell transplantation
* Presence of co-morbidities (hematopoietic cell transplant co-morbidity index [HCT-CI] score 3 or greater), high risk disease (relapse risk > 25%), or a planned type of transplant (human leukocyte antigen [HLA]-mismatched allogeneic or myeloablative) that places the patient at a higher than average risk of non-relapse mortality or relapse

Exclusion Criteria:

* Major psychiatric diagnosis that impairs cognitive functioning or is not controlled at the time of the approach, as judged by the patient's medical team
* First transplant of a planned tandem procedure (the second transplant is eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Study participation rates defined as the proportion of patients who consent to enroll | Up to 5 months
  Will mainly be descriptive.
Completion time for the supportive care consultation | Up to 90 days post-treatment
  Will mainly be descriptive.
Level of comfort / distress attributed to individual parts of the consultation | Up to 90 days post-treatment
  Will mainly be descriptive. The post-consultation scores measuring level of comfort or distress per topic in the supportive care consultation will be summarized per item.
Completeness of follow-up data collection, where completeness is defined by the proportion of instrument scores that can be calculated per given time point | Up to 90 days post-treatment
  Will mainly be descriptive. The completeness of follow-up data collection will be calculated and reported as a proportion of successfully completed scales vs. scales attempted to be collected or completed by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States